CLINICAL TRIAL: NCT04042597
Title: A Prospective, Multicentre, Open-label, Randomised Phase 2 Trial to Study the Efficacy and Safety of Anlotinib Hydrochloride Versus Imatinib Mesylate in Locally Advanced, Unresectable or Metastatic Chordoma
Brief Title: Anlotinib Hydrochloride Versus Imatinib Mesylate in Locally Advanced, Unresectable or Metastatic Chordoma
Acronym: CSSG-03
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Peking University Third Hospital (Other); Peking University First Hospital (Other); Beijing Jishuitan Hospital (Other); Chinese PLA General Hospital (Other); Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 05
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Effect of Drugs; Quality of Life; Chordoma; Advanced Cancer
Keywords: chordoma; unresectable; anlotinib; imatinib; survival; quality of life
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: anlotinib arm (Experimental): anlotinib was given at a fixed dose of 12mg D1-14 every 21 days
  Interventions: Drug: Anlotinib Hydrochloride
- Arm B: imatinib arm (Active Comparator): Imatinib was given at dose of 400 mg twice daily continuously
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — anlotinib was given at a fixed dose of 12mg D1-14 every 21 days

SUMMARY:
For local relapse not amenable to reasonable curative surgery or for those with metastatic chordoma, chemotherapy is recognised as inactive. The major study drug is the small molecular tyrosine kinase inhibitors targeted at the stem cell factor receptor (KIT) and the platelet-derived growth factor receptors (PDGFRA and PDGFRB), eg. imatinib. Anlotinib is a novel tyrosine kinase inhibitor targeting both at VEGFR-2, -3 and PDGFRA and PDGFRB with high affinity, which also showed broad antitumor activity against EGFR and so on. Thus this multicenter, two-armed phase II trial of PKUPH-sarcoma 05 intended to investigate the efficacy and safety of anlotinib versus imatinib on advanced chordoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older;
* histologically proven metastatic or locally advanced chordoma, reviewed by the Pathology Committee of Peking University People's Hospital;
* not amenable to curative-intent surgery;
* measurable with computed tomography scan or magnetic resonance imaging, per RECIST, version 1.1.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG)30 performance status more than 2 ;
* life expectancy less than 12 weeks;
* with severe or uncontrolled medical disorders (≥grade 2 of Common Terminology Criteria for Adverse Events version 4.03 [CTCAE version 4.03]) that could jeopardise the outcomes of the study, for example, cardiac clinical symptom or disease with LVEF (left ventricular ejection fraction) <50%, hypertension that could not be well controlled through antihypertensive drugs and so on;
* weight loss of 20% or more before illness;
* brain or leptomeningeal metastasis;
* surgical procedure or radiotherapy within 4 weeks of enrollment;
* active gastroduodenal ulcer, previous condition associated with risk of bleeding or requiring anticoagulation;
* proteinuria or hematuria;
* denutrition with albuminemia less than 25 g/L;
* pregnant or breastfeeding status;
* other malignancy, positive HBV/HCV/HIV serology;
* known allergy to the experimental agents;
* had ever used anti-angiogenesis TKIs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 6 months
  CR+PR in the intent-to-treat population according to RECIST, version 1.1
Progression-free Survival, PFS | 2 years
  Progression-free survival is defined as time from randomisation to the first occurrence of progression of disease or death from any cause within 63 days of last response assessment or randomisation

SECONDARY OUTCOMES:
Overall Survival, OS | 5 years
  OS is defined as time from randomisation to the first occurrence of death from any cause within 63 days of last response assessment or randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D. and Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No